CLINICAL TRIAL: NCT06772311
Title: Clinical Efficacy of Surgical Vs. Conservative Treatment for Atlantoaxial Dislocation Patients Without Neurological Deficit: a Prospective, Multicenter, Observational Study
Brief Title: Conservative Treatment for Atlantoaxial Dislocation Patients Without Neurological Deficit
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Shanxi Medical University Second Hospital (Unknown); Sir Run Run Shaw Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Hebei Medical University Third Hospital (Other); Shanxi Bethune Hospital (Other); Daping Hospital of Army Medical University (Other); Shengjing Hospital (Other); Tianjin People's Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Affiliated hospital of Guilin medical university,China (Unknown)
Responsible Party: Principal Investigator, Wang Shenglin, Professor, Peking University Third Hospital
Other Study IDs: M20248745
Record Dates: First submitted 2025-01-01; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Atlantoaxial Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No samples will be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conservative Treatment Group: Patients who declined surgery and request conservative treatment and observation.
- Surgical Intervention Group: Patients who request surgical intervention.

SUMMARY:
The goal of this observational study was to learn about the long-term clinical efficacy of conservative treatment in atlantoaxial dislocation patients without neurological deficit. The main question it aims to answer is:

Is surgical intervention always necessary in atlantoaxial dislocation patients without nerve deficit?

Patients who refuse surgical intervention will continue to be treated conservatively. Clinical outcomes will be summarized over five years of follow-up

ELIGIBILITY:
Inclusion Criteria:

* The patients meet the diagnostic criteria for atlantoaxial dislocation, that is, the ADI exceeds the normal range: it is over 3 mm in adults and over 5 mm in children.
* The patients have no clinical manifestations of the nervous system, including occipital neuralgia, manifestations of cranial nerve impairment (such as dysphagia, dysarthria, nystagmus, etc.) and manifestations of spinal cord impairment (such as unsteadiness in holding objects, unsteady gait, decreased limb muscle strength, etc.).
* After fully understanding their own conditions as well as the advantages, disadvantages and risks of both conservative treatment and surgical treatment, the patients can choose the initial treatment method on their own. If they choose conservative treatment, they will be included in the conservative treatment. If they choose surgical treatment, they will be included in the surgical intervention group.

Exclusion Criteria:

* Patients who have undergone surgeries in the cranio-cervical junction previously.
* Patients with infections or tumors in the cranio-cervical junction.
* Patients with fresh fractures in the cranio-cervical junction.
* Patients with clinical manifestations of nerve deficit.
* Patients with severe diseases in other spinal regions such as the thoracic and lumbar spine that affect their clinical symptoms; patients with motor neuron diseases like amyotrophic lateral sclerosis and other severe neurological diseases.
* Patients who have participated in other clinical trials within the recent three months.
* Patients with mental disorders whose cognitive impairments (or those of their legal guardians) prevent them from giving full informed consent.
* Patients who refuse to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Atlantoaxial dislocation patients without neurological deficit.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of neurological deficit | The incidence of neurological deficit will be assessed at the initial visit, and at 3 months, 6 months, and 12 months after the initial visit, with annual follow-ups thereafter. Follow-up will continue for at least 5 years.
  The incidence of neurological deficit is defined as the proportion of patients with neurological deficit to the total number of patients during the research period. Neurological deficit includes cranial nerve involvement and spinal cord involvement, with specific clinical manifestations such as occipital neuralgia, dysphagia, dysarthria, nystagmus, unsteadiness in holding objects, unsteady gait, decreased limb muscle strength, paralysis, and others.

SECONDARY OUTCOMES:
Japanese Orthopaedic Association score | The JOA score will be assessed at the initial visit, and at 3 months, 6 months, and 12 months after the initial visit, with annual follow-ups thereafter. Follow-up will continue for at least 5 years.
  The Japanese Orthopaedic Association (JOA) score is a widely used disease-specific outcome tool that can provide a quantitative measure for patients with cervical myelopathy. JOA score consists of 6 domains: motor function in upper extremities, motor function in lower extremities, sensory function in upper extremities, sensory function in the trunk, sensory function in lower extremities, and bladder function, with a minimum total score of 0 and maximum of 17.
Neck Disability Index | The NDI will be assessed at the initial visit, and at 3 months, 6 months, and 12 months after the initial visit, with annual follow-ups thereafter. Follow-up will continue for at least 5 years.
  The Neck Disability Index (NDI) is the most widely used assessment tool measuring disability due to neck pain or neck injury. The NDI consists of 10 items: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The total score for the NDI is out of 50. A higher total score indicates a higher level of disability.
ADI | The ADI will be assessed at the initial visit, and at 3 months, 6 months, and 12 months after the initial visit, with annual follow-ups thereafter. Follow-up will continue for at least 5 years.
  Atlantodental Interval (ADI) refers to the distance between the anterior tubercle of the atlas and the odontoid process, which reflects the severity of atlantoaxial dislocation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No